CLINICAL TRIAL: NCT01124019
Title: SNP Panels and Risk Assessment in Women Undergoing Mammography
Brief Title: Single Nucleotide Polymorphism (SNP) Panels and Risk Assessment in Women Undergoing Mammography
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 17109
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Mammography
Keywords: Women undergoing screening mammography will be chosen if they are between the ages of 40 and 65.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Random Sample: A random sample of 600 women undergoing screening mammography
- BIRADS score of 4: An additional 600 women determined to have a Breast Imaging Reporting and Data System (BIRADS) score of 4 as determined by final mammogram results.

SUMMARY:
The primary objective is to compare the predicted lifetime risk values produced by SNP panel assessment to the risk values produced by the prediction models that are most commonly used. A second objective is to examine whether the incorporation of risk assessment panels (standard or SNP based) can improve the positive value of breast biopsies in women with BIRADS 4 mammograms.

DETAILED DESCRIPTION:
Calculating the risk that a woman will develop breast cancer in her lifetime can lead to decreased mortality rates as a result of increased screening and prevention methods when a person is known to be at high risk. Though there are several risk assessment models that are commonly used, it is important to continue to improve the process of calculating risk. Several genetic markers have been noted to potentially indicate risk of developing breast cancer. New tests, called SNP panels, can detect some of these genetic markers. This study aims to use both these SNP panels and the commonly used risk models to calculate risk and examine outcomes in women coming in to do screening mammography. This study will enroll women between the ages of 40-65 who are undergoing screening mammography (n=1000), in addition to women with BIRADS category 4 mammogram readings who are about to undergo biopsy (n=600), all with no personal history of breast or ovarian cancer, ductal carcinoma in situ (DCIS), mantle radiation, or known BRCA 1/2/mutation in self or family members. The participants will only be expected rto provide consent, swabs of the inside of the cheek of her mouth, and baseline questionnaire answers that will allow for a risk assessment to be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 40 and 65 years old undergoing screening mammography at the University of Pennsylvania Health System and women undergoing biopsy as the result of a BIRADS category 4 mammogram result.

Exclusion Criteria:

* Women will be excluded if they have a personal history of breast or ovarian cancer, DCIS, or mantle radiation, or known BRCA 1/2 mutation in self or in family members.
* In addition, women younger than 40 or older than 65 will be excluded if they are in the screening mammography population of potential participants.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women will be recruited for this study. Women undergoing screening mammography will be chosen if they are between the ages of 40 and 65. Women will be excluded if they have a personal history of breast or ovarian cancer, DCIS, or mantle radiation, or known BRCA 1/2 mutation in self or in family members.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Predicted Risk Category and Prevention Recommendations
  The predicted risk category and prevention recommendations which are based upon the category each patient falls into after risk assessment using either a traditional or a SNP-based approach. Change in PPV of mannographic biopsy by stratification into low and high risk groups.

SECONDARY OUTCOMES:
Tests and Evaluations
  Secondary Outcome will be determining the number of women who are ordered and/or complete tests and/or evaluations if there are abnormal imaging results during mammography or if they have high lifetime risk. These will be measured through access to the electronic medical records (EMR) and/or through a follow up survey.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States